CLINICAL TRIAL: NCT02223936
Title: Follow up of Neurologic Development of Children Who Presented at the First Trimester of Pregnancy an Isolated Nuchal Anomaly With Normal Karyotype
Acronym: EDEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2007-491
Record Dates: First submitted 2014-08-12; First posted 2014-08-22 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-07

CONDITIONS: Neurological Development After Exposition to an Antenatal Nuchal Translucency
Keywords: nuchal translucency, neurological developpment, anxiety, depression, prenatal diagnosis, normal karyotype
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- children with Prenatal enlarged nuchal transluce (Other)
  Interventions: Other: group exposed
- Control (Other)
  Interventions: Other: Control

INTERVENTIONS:
Other: group exposed — Assessment by Brunet Lezine scale
  Arms: children with Prenatal enlarged nuchal transluce
Other: Control — Not exposed group
  Arms: Control

SUMMARY:
Prospective, multicenter study following for 2 years, 250 children who presented during the first trimester of pregnancy an isolated nuchal translucency over the 95th percentile of Nicolaïdes Curves on ultrasound and comparing them to a control group of 250 children whose pregnancy was normal. Evaluating morbidity, mortality, growth and the neurodevelopment of each group by a Brunet Lezine scale. Evaluating anxiety and depression in parents of those children using a scale.

ELIGIBILITY:
Inclusion Criteria:

-

Confirmation of the enlargement of nuchal tranlucency by a sonographer referent OR ultrasound abnormality neck restraint by sonographers referents replay after the initial shots (the notion of transience of the pathology of the neck being allowed) with in all cases:

* gestational age between 11 and SA 13 SA 0 days 6 days or a crown-rump length between 45 and 84 mm
* Thickness of the neck> 95th percentile of the standard set for the crown-rump length according to the team Nicolaides
* ultrasound Clichés meet quality criteria HERMANN (score ≥ 5 at least 2 major criteria).
* normal karyotype or not done
* Morphological Ultrasound second quarter normal or minor abnormalities

  * Consent signed holders of parental authority for monitoring up to 2 years and neurodevelopmental assessment at the end of follow-up
  * Affiliate or benefit of a social security scheme.

Exclusion Criteria:

* Multiple Pregnancy

  * Prematurity less than 32 SA
  * Birth weight less than 1500 grams
  * Discovery of a chromosomal abnormality on karyotype not made prenatally
  * Withdrawal of consent.
  * intercurrent Event may be the cause of abnormal psychomotor development: fetal distress cause of hospitalization, prenatal viral infection

Inclusion Criteria: for control group

* Newborn who did not have enlarged nuchal translucency and with normal antenatal ultrasound.
* Matching each child the "nuchal group" on:

  * Maternity Birth: matching the child witness in the University Hospital of the same region as motherhood in which the child with nuchal group is born.
  * gestational age: the child matched group must belong to the same group of gestational age than neck the child with nuchal group

    * ≥ 37 weeks
    * ≥ 32 and <37 weeks with a less than 2 SA difference
  * Weight:

    * if the weight of the child of nuchal group is ≥ 2500g, the weight of the child must also be matched to ≥ 2500g and with a weight difference between the two children ≤ 500g
    * If the weight of the child of nuchal group is ≥ 1500g and less than 2500g, the weight of the child must also be matched to ≥ 1500g and less than 2500 g and with a weight difference between the two children ≤ 200g
  * Apgar score at 5 minutes: the difference in Apgar score at 5 minutes between the two children should be zero or at most equal to 1
  * birth: same according to the following criteria:

    * primipara
    * Multiparous
* Consent signed holders of parental authority for neurodevelopmental assessment and monitoring at the age of 2 years.
* Children with no 21 trisomy, or other intercurrent disease may be responsible for neurodevelopmental

Max Age: 26 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Actual)
Dates: Start 2009-02; Primary Completion 2011-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Incidence of developmental quotient below 70 compared to a group control | Assessment at the age of 2 years + / - 45 days for each patient
  assessed by the Brunet Lezine test

SECONDARY OUTCOMES:
comparison of the mean and distribution of developmental quotient between the two arms | at the age of 2 years + / - 45 days
  assessed by the Brunet Lezine test
composite outcome measure : comparison of weight, height and head circumference between the two arms | at 3 months, 1 year and 2 years
  assessed by measurement
The status deceased / living and the date and cause of death if applicable | any time after birth and before 2 years + / - 45 days
  nterview
study differences in score post-traumatic stress, anxiety and depression between parents of the two arms | at the consultation at the age of 2 years + / - 45 days of the children
  assessment of the questionnaire of posttraumatic stress and HAD scale by the parents during the consultation of the two-year child

CONTACTS AND LOCATIONS:
Overall Officials: Rachel BUFFIN, Dr, Study Director — Hospices Civils de Lyon